CLINICAL TRIAL: NCT01897597
Title: An Open-label, Single Dose, Randomised, Crossover Trial in Healthy Male Subjects to Investigate the Relative Bioavailability of Tablet and Oral Solution of Two Doses of BI 144807 and Relative Bioavailability of BI 144807 When Administered as Tablet Under Fed and Fasted Conditions
Brief Title: Clinical Drug Trial in Healthy Male Subjects to Determine and Compare the Blood Concentrations of BI 144807 Following Administration as Oral Solution and Tablet Under Fasted and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1313.9; 2013-000258-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Healthy

ARMS (7):
- BI 144807 PfoS Treatment A (Experimental): intermediate dose of BI 144807
  Interventions: Drug: BI 144807 intermediate dose
- BI 144807 PfoS Treatment C (Experimental): high dose of BI 144807
  Interventions: Drug: BI 144807 high dose
- BI 144807 Tab Treatment B (Experimental): intermediate dose of BI 144807
  Interventions: Drug: BI 144807 intermediate dose
- BI 144807 Tab Treatment D (Experimental): high dose of BI 144807
  Interventions: Drug: BI 144807 high dose
- BI 144807 Tab Treatment E (Experimental): intermediate dose of BI 144807, fasted
  Interventions: Drug: BI 144807 intermediate dose
- BI 144807 Tab Treatment F (Experimental): intermediate dose of BI 144807, fed
  Interventions: Drug: BI 144807 intermediate dose
- BI 144807 Tab Treatment G (Experimental): intermediate dose of BI 144807, fasted
  Interventions: Drug: BI 144807 intermediate dose

INTERVENTIONS:
Drug: BI 144807 high dose — oral solution
  Arms: BI 144807 PfoS Treatment C
Drug: BI 144807 intermediate dose — tablet
  Arms: BI 144807 Tab Treatment F
Drug: BI 144807 intermediate dose — tablet
  Arms: BI 144807 Tab Treatment E
Drug: BI 144807 intermediate dose — tablet
  Arms: BI 144807 Tab Treatment G
Drug: BI 144807 intermediate dose — tablet
  Arms: BI 144807 Tab Treatment B
Drug: BI 144807 intermediate dose — oral solution
  Arms: BI 144807 PfoS Treatment A
Drug: BI 144807 high dose — tablet
  Arms: BI 144807 Tab Treatment D

SUMMARY:
The purpose of this trial is to investigate the relative bioavailability of a BI 144807 tablet formulation compared to the oral solution formulation after single dose administration (intermediate and high dose) under fasted conditions. Further objectives are to assess whether and to what extent food affects single dose pharmacokinetics of BI 144807 administered as tablet, and to compare the relative bioavailability of two different tablet formulations.

ELIGIBILITY:
Inclusion criteria:

- Healthy male subjects

Exclusion criteria:

- Any relevant deviation from healthy condition

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | 48 hours
Maximum measured concentration of the analyte in plasma (Cmax) | 48 hours

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1313.9.1 Boehringer Ingelheim Investigational Site, Biberach, Germany